CLINICAL TRIAL: NCT01416389
Title: A Randomized Phase 2 Study of LY2523355 Versus Ixabepilone in Patients With Metastatic or Locally Recurrent Breast Cancer Who Have Received Prior Taxane Therapy
Brief Title: A Study of LY2523355 in Participants With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12847; I1Y-MC-JFBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Locally; Recurrent; Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasms | interventions — litronesib; ixabepilone; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2523355 + pegfilgrastim or filgrastim (Experimental): LY2523355: Five milligrams per meter squared per day (mg/m^2/day) (dosage determined by calculating participant's body surface area) administered intravenously as a 1-hour infusion on Days 1, 2, and 3 of a 21-day Cycle for 2 Cycles. Pegfilgrastim or Filgrastim: Dosage is determined by standard of care and is administered intravenously on Day 4 of 21-day Cycle for 2 Cycles. If at the end of 2 Cycles the participant was receiving benefit, the participant may have remained on study drug for additional cycles until a criterion for study discontinuation was met.
  Interventions: Drug: LY2523355; Drug: pegfilgrastim; Drug: filgrastim
- ixabepilone (Active Comparator): Forty milligrams per meter squared per day (mg/m^2/day) (dosage determined by calculating participant's body surface area) administered intravenously as a 3-hour infusion on Day 1 of a 21-day Cycle for 2 Cycles. If at the end of 2 Cycles the participant was receiving benefit, the participant may have remained on study drug for additional cycles until a criterion for study discontinuation was met.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: LY2523355 — Administered intravenously as a one hour infusion
  Arms: LY2523355 + pegfilgrastim or filgrastim
Drug: ixabepilone — Administered intravenously
  Arms: ixabepilone
Drug: pegfilgrastim — Administered intravenously
  Arms: LY2523355 + pegfilgrastim or filgrastim
Drug: filgrastim — Administered intravenously
  Arms: LY2523355 + pegfilgrastim or filgrastim

SUMMARY:
The purpose of the study is to evaluate the anti-tumor activity of LY2523355 relative to ixabepilone for the treatment of metastatic or locally recurrent breast cancer using change in tumor size as a continuous measure of response.

ELIGIBILITY:
Inclusion Criteria:

* Have histologic or cytologic diagnosis of metastatic or locally recurrent breast cancer that is not amenable to therapy given with curative intent.
* Have measurable disease defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 guidelines.
* Have received 2 or more prior standard cytotoxic chemotherapy regimens for metastatic breast cancer and be, in the opinion of the investigator, an appropriate candidate for experimental therapy. Regimens received in the neoadjuvant or adjuvant setting are not counted as prior regimens.
* Have received a prior taxane in the neoadjuvant, adjuvant, or metastatic setting.
* Have recovered from the acute effects of prior chemotherapy, hormonal therapy, and radiation prior to study enrollment.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have adequate organ function.

Exclusion Criteria:

* Have Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater (moderate or worse) peripheral neuropathy
* Have a second primary malignancy.
* Have symptomatic, untreated, or uncontrolled central nervous system metastases.
* Have received autologous stem cell transplant following high-dose chemotherapy.
* Have serious preexisting medical conditions that in the opinion of the investigator would preclude participation in this study.
* Have active symptomatic fungal, bacterial, and/or known viral infection including active human immunodeficiency virus (HIV) or viral hepatitis.
* Have previously received LY2523355 in another study investigating this agent or therapy with ixabepilone or an ixabepilone-containing regimen.
* Have a history of radiation therapy involving more than 25 percent of the bone marrow.
* Have a Fridericia corrected QT (QTcF) interval of >470 milliseconds (msec) on screening electrocardiogram (ECG).
* Have QRS widening of >120 msec on screening ECG.
* Cannot change or stop taking a strong Cytochrome P450 3A4 (CYP3A4) inhibitor or CYP3A4 inducer per the ixabepilone label.
* Have hypersensitivity to drugs formulated with Cremophor® EL per the ixabepilone label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hour, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pensacola, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spartanburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the study if they had at least 1 dose of study drug in Cycle 2 (or later) and had at least 1 post-baseline radiological tumor assessment or if the participant had a progression of disease or death. Non-completers were those that were lost to follow-up or who withdrew their consent to trial participation.
Groups:
- LY2523355 + Pegfilgrastim or Filgrastim: LY2523355 administered intravenously as a 1-hour infusion on Days 1, 2, and 3 of a 21-day Cycle for 2 Cycles. Dosage determined by calculating participant's body surface area (5 milligrams per meter squared per day [mg/m^2/day]). One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2. The dose was subsequently corrected and the participant is included in this analysis.
  Pegfilgrastim or filgrastim administered intravenously on Day 4 of 21-day Cycle for 2 Cycles. Dosage is determined by standard of care.
  If at the end of 2 Cycles the participant was receiving benefit, the participant may have remained on study drug for additional cycles until a criterion for study discontinuation was met.
- Ixabepilone: Ixabepilone administered intravenously as a 3-hour infusion on Day 1 of a 21-day Cycle for 2 Cycles.
  Dosage determined by calculating participant's body surface area (40 mg/m^2).
  If at the end of 2 Cycles the participant was receiving benefit, the participant may have remained on study drug for additional cycles until a criterion for study discontinuation was met.
Period: Overall Study
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Started | 26 | 13
Received at Least 1 Dose of Study Drug | 26 | 13
Completed | 23 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Started New Therapy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study medication (LY2523355 or ixabepilone). One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2. The dose was subsequently corrected and the participant is included in this analysis.
Groups:
- LY2523355 + Pegfilgrastim or Filgrastim: LY2523355 administered intravenously as a 1-hour infusion on Days 1, 2, and 3 of a 21-day Cycle for 2 Cycles. Dosage determined by calculating participant's body surface area (5 milligrams per meter squared per day [mg/m^2/day]).
  Pegfilgrastim or filgrastim administered intravenously on Day 4 of 21-day Cycle for 2 Cycles. Dosage is determined by standard of care.
  If at the end of 2 Cycles the participant was receiving benefit, the participant may have remained on study drug for additional cycles until a criterion for study discontinuation was met.
- Total: Total of all reporting groups
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.9) | 57.8 (9.9) | 60.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 13 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 13 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 21 | 9 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Size (CTS) From Baseline to the End of Cycle 2
Description: The log ratio of tumor size at Cycle 2 to tumor size at baseline is calculated for each participant, where the tumor size is the sum of the target lesion measurements at each assessment.
Time Frame: Baseline up to end of Cycle 2 (Day 42)
Population: Participants who received at least 1 dose of study medication (LY2523355 or ixabepilone) and who had target lesion measurements at both baseline and the end of Cycle 2. One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2. The dose was subsequently corrected and the participant is included in this analysis.
Measure: Mean (Standard Deviation); unit: log ratio of end of Cycle 2 to baseline
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Number analyzed (Participants) | 17 | 11
log ratio of end of Cycle 2 to baseline | -0.0 (0.08) | -0.1 (0.37)
Statistical Analysis 1: Comparison: LY2523355 + Pegfilgrastim or Filgrastim vs Ixabepilone; This measure is compared between two treatment arms using a one-sided t-test. This measure followed a normal distribution; Test type: Superiority or Other; p = 0.344, t-test, 1 sided

2. Secondary Outcome: Percentage of Participants Achieving an Overall Response (Overall Response Rate)
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guidelines. CR is a disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). PR is an at least 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with measurable disease, multiplied by 100.
Time Frame: Baseline to measured progressive disease or date of death from any cause (up to 423 days)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of responders
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Number analyzed (Participants) | 26 | 13
percentage of responders | 3.8 [0.2 to 17] | 7.7 [0.4 to 31.6]
Statistical Analysis 1: Comparison: LY2523355 + Pegfilgrastim or Filgrastim vs Ixabepilone; Test type: Superiority or Other; p = 0.608, Chi-squared

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is the time from the date of randomization to the first date of progressive disease (PD) or death due to any cause, whichever occurs first. PD is as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guidelines, and is defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if that was the smallest on study). In addition, the sum must have demonstrated an absolute increase of at least 5 millimeter (mm) (the appearance of 1 or more new lesions was considered progression). Kaplan-Meier analysis was performed on the observed distribution of PFS. Participants were censored from analysis for the following reasons: lack of disease assessment, lost to follow-up, and further anticancer therapy started. Median PFS is presented.
Time Frame: Baseline to measured progressive disease or date of death from any cause (up to 423 days)
Population: Participants who received at least 1 dose of study medication (LY2523355 or ixabepilone). The total number of participants censored is 7. One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2. The dose was subsequently corrected and the participant is included in this analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Number analyzed (Participants) | 22 | 10
months | 1.71 [1.25 to 2.79] | 2.76 [1.41 to 4.80]

4. Secondary Outcome: Percentage of Participants Achieving a Clinical Benefit (Clinical Benefit Rate)
Description: Clinical benefit rate is the proportion of participants who achieve a best response of complete response (CR), partial response (PR), or stable disease (SD) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guidelines. CR is a disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). PR is an at least 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. SD is neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as progressive disease, taking as reference the smallest sum diameter since treatment started.
  Clinical benefit rate is calculated as a total number of participants with CR, PR, or SD divided by the total number of participants with measurable disease, multiplied by 100.
Time Frame: Baseline to measured progressive disease or date of death from any cause (up to 423 days)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of responders
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Number analyzed (Participants) | 26 | 13
percentage of responders | 46.2 [29.2 to 63.8] | 61.5 [35.5 to 83.4]
Statistical Analysis 1: Comparison: LY2523355 + Pegfilgrastim or Filgrastim vs Ixabepilone; Test type: Superiority or Other; p = 0.365, Chi-squared

5. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax) of LY2523355
Description: Cmax is the maximum plasma concentration of LY2523355 after a 1-hour intravenous infusion of LY2523355 on Day 1 and Day 3 of Cycle 1.
Time Frame: Cycle 1: Day 1 and Day 3
Population: Participants who received 1 dose of LY2523355 on Day 1 and Day 3 of Cycle 1 and who have evaluable pharmacokinetic data to enable estimation of the LY2523355 Cmax on Day 1 and Day 3 of Cycle 1. One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2, and is not included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- LY2523355: LY2523355 administered intravenously as a 1-hour infusion on Days 1, 2, and 3 of a 21-day Cycle for 2 Cycles. Dosage determined by calculating participant's body surface area (5 milligrams per meter squared per day [mg/m^2/day]).
Arm/Group | LY2523355
Number analyzed (Participants) | 24
nanograms/milliliter (ng/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 21
  Cycle 1, Day 1 | 161 (81)
  Cycle 1, Day 3 | 150 (56)

6. Other Pre Specified Outcome: Percentage of Deaths on Study Through the Follow-up Period
Description: The percentage of participants who died through the follow-up period of the study; the cause of death was not captured.
  A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through end of treatment follow-up (up to 423 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Number analyzed (Participants) | 26 | 13
percentage of participants | 7.7 | 15.4

7. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax) of LSN2546307
Description: Cmax is the maximum plasma concentration of LSN2546307 (metabolite) after a 1-hour intravenous infusion of LY2523355 on Day 1 and Day 3 of Cycle 1.
Time Frame: Cycle 1: Day 1 and Day 3
Population: Participants who received 1 dose of LY2523355 on Day 1 and Day 3 of Cycle 1 and who have evaluable pharmacokinetic data to enable estimation of the LSN2546307 Cmax on Day 1 and Day 3 of Cycle 1.One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2, and is not included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- LSN2546307: LSN2546307 is the metabolite of LY2523355. LY2523355 administered intravenously as a 1-hour infusion on Days 1, 2, and 3 of a 21-day Cycle for 2 Cycles. Dosage determined by calculating participant's body surface area (5 milligrams per meter squared per day [mg/m^2/day]).
Arm/Group | LSN2546307
Number analyzed (Participants) | 24
nanograms/milliliter (ng/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 21
  Cycle 1, Day 1 | 5.08 (57)
  Cycle1, Day 3 | 5.53 (67)

8. Secondary Outcome: Pharmacokinetics, Intracycle Accumulation Ration (Ra) of LY2523355
Description: The intracycle accumulation ratio (Ra) is defined as the LY2523355 Cmax on Day 3 of Cycle 1 to the LY2523355 Cmax on Day 1 of Cycle 1 after a 1-hour intravenous infusion of LY2523355 on Day 1 and Day 3 of Cycle 1.
Time Frame: Cycle 1: Day 1 and Day 3
Population: Participants who received 1-dose of LY2523355 on Day 1 and Day 3 of Cycle 1 and who have evaluable pharmacokinetic data to enable estimation of the LY2523355 Cmax on Day 1 and Day 3 of Cycle 1. One participant was mistakenly dosed with 6 mg/m^2/day in Cycle 1 and for 2 doses in Cycle 2, and is not included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: unitless ratio
Arm/Group | LY2523355
Number analyzed (Participants) | 21
unitless ratio | 0.92 (77)

ADVERSE EVENTS:
Arm/Group | LY2523355 + Pegfilgrastim or Filgrastim | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 5/26 | 4/13
Other Adverse Events (participants affected / at risk) | 26/26 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2523355 + Pegfilgrastim or Filgrastim (N=26) | Ixabepilone (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2523355 + Pegfilgrastim or Filgrastim (N=26) | Ixabepilone (N=13)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 5 (5)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (13) | 5 (5)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (1)
Globulins decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days